CLINICAL TRIAL: NCT03385811
Title: Exploring the Correlation of ProQOL, Health Status, Job Involvement, Intention to Stay and Turnover Behaviour in Medical Professionals
Brief Title: Exploring ProQOL, Health Status, Job Involvement and Turnover in Medical Professionals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Li-chi Huang, associate professor, China Medical University Hospital
Other Study IDs: CRREC-106-085
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-11

CONDITIONS: Intention to Stay, Turnover Behavior
Keywords: Professional quality of life, Medical Professionals, Job Involvement, Intention to Stay,

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical Professionals: no intervention, only questionnaire survey
  Interventions: Other: no intervention, only questionnaires survey

INTERVENTIONS:
Other: no intervention, only questionnaires survey — questionnaires survey
  Other Names: no intervention

SUMMARY:
The study design is a cross-sectional study. Purposive sampling will be conducted in three hospitals in the central of Taiwan. The participants will include physicians, nurse practitioners and nurses. The number of 550 participants will be recruited. The measurements are questionnaires include demographic data, professional quality of life scale (ProQOL), Job Involvement Questionnaire (JIQ), SF-36 and intention to stay questionnaire.

DETAILED DESCRIPTION:
Medical and Nursing care is a high-pressure work environment. The charterer of medical and nursing care includes urgency of patients' problems, an unpredictable number of patients, and lack of medical professionals. This high-level of pressure working environment not only affects the persons' physical and mental health, increase turnover rate, but also might indirectly reduce the quality of care, even threaten the life of patients.

The purpose of this study is to explore the correlation between professional quality of life, health status, job involvement and intention to stay in medical professionals, and the predictive factors of intention to stay and turnover behavior.

The study design is a cross-sectional study. Purposive sampling will be conducted in three hospitals in the central of Taiwan. The participants will include physicians, nurse practitioners, and nurses. The number of 550 participants will be recruited. The measurements are questionnaires include demographic data, professional quality of life scale (ProQOL), Job Involvement Questionnaire (JIQ), SF-36 and intention to stay questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 20 years old
2. Currently serving as a hospital care provider
3. Job title as attending physician, resident, nurse practitioners, nurse
4. Directly practicing in patients' care

Exclusion Criteria:

1. Medical Director
2. Clinical Researcher

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical professions who work in the hospital
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
professional quality of life scale | within past 30 days
  Professional quality of life scale consists of compassion satisfaction (CS), burnout(BO), and secondary traumatic stress (compassion fatigue, CF)
Job Involvement Questionnaire (JIQ) | within past 30 days
  Job Involvement Questionnaire (JIQ) includes 4 items
SF-36 | within past 30 days
  36 items
intention to stay questionnaire | within past 30 days
  6 items

CONTACTS AND LOCATIONS:
Overall Officials: Li-Chi Huang, Study Chair — Associate Professor, Nursing school, China Medical Univerisity, Taiwan.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mason VM, Leslie G, Clark K, Lyons P, Walke E, Butler C, Griffin M. Compassion fatigue, moral distress, and work engagement in surgical intensive care unit trauma nurses: a pilot study. Dimens Crit Care Nurs. 2014 Jul-Aug;33(4):215-25. doi: 10.1097/DCC.0000000000000056. PMID 24895952
- [Result] Neville K, Cole DA. The relationships among health promotion behaviors, compassion fatigue, burnout, and compassion satisfaction in nurses practicing in a community medical center. J Nurs Adm. 2013 Jun;43(6):348-54. doi: 10.1097/NNA.0b013e3182942c23. PMID 23708503
- [Result] Bellolio MF, Cabrera D, Sadosty AT, Hess EP, Campbell RL, Lohse CM, Sunga KL. Compassion fatigue is similar in emergency medicine residents compared to other medical and surgical specialties. West J Emerg Med. 2014 Sep;15(6):629-35. doi: 10.5811/westjem.2014.5.21624. PMID 25247031
- [Result] Hinderer KA, VonRueden KT, Friedmann E, McQuillan KA, Gilmore R, Kramer B, Murray M. Burnout, compassion fatigue, compassion satisfaction, and secondary traumatic stress in trauma nurses. J Trauma Nurs. 2014 Jul-Aug;21(4):160-9. doi: 10.1097/JTN.0000000000000055. PMID 25023839
- [Result] Hunsaker S, Chen HC, Maughan D, Heaston S. Factors that influence the development of compassion fatigue, burnout, and compassion satisfaction in emergency department nurses. J Nurs Scholarsh. 2015 Mar;47(2):186-94. doi: 10.1111/jnu.12122. Epub 2015 Jan 20. PMID 25644276